CLINICAL TRIAL: NCT07100925
Title: An Open-Label Study of Tolododekin Alfa (ANK-101) in Renal Allograft Recipients With Resectable, High-Risk Cutaneous Squamous Cell Carcinoma
Brief Title: A Study of Tolododekin Alfa (ANK-101) in Renal Allograft Recipients With High Risk Cutaneous Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ankyra Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANK-101-003
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Cutaneous Squamous Cell Carcinoma (CSCC); Renal Transplant; Solid Tumor; Solid Tumor Cancer
Keywords: intratumoral injection; intratumoral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- tolododekin alfa (ANK-101) IT Injection (Experimental): Participants will receive 2 cycles of tolododekin alfa before surgical resection of CSCC tumor
  Interventions: Drug: tolododekin alfa

INTERVENTIONS:
Drug: tolododekin alfa — IT administration of ANK-101 once every 3 weeks for 2 cycles, followed by surgical resection

SUMMARY:
A study of tolododekin alfa (also known as ANK-101) administered prior to surgery in kidney transplant participants that also have high-risk cutaneous squamous cell carcinoma (CSCC).

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed high-risk and/or locoregionally metastatic CSCC
2. Have measurable disease per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
3. Are renal allograft recipients on a stable immunosuppressive regimen.
4. Have adequate renal function defined as creatinine clearance ≥ 30 mL/min as determined by the Cockcroft-Gault equation.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
6. Have a life expectancy > 12 months.
7. Have baseline electrocardiogram (EKG) without evidence of acute ischemia or prolonged QT interval
8. Heterosexually active women of childbearing potential (WOCBP) must agree to use at least 2 forms of highly effective methods of contraception
9. All male participants who are not sterile must commit to the use of a reliable method of birth control or abstinence.
10. Last dose of previous anticancer therapy (including investigational agents) ≥ 28 days or surgical intervention ≥ 21 days prior to the first dose of study drug.
11. Resolution of all prior anticancer therapy toxicities (except for alopecia or vitiligo) to ≤ Grade 1
12. Willingness to provide fresh tumor biopsy specimens
13. Capable of understanding and complying with protocol requirements.
14. Provides written informed consent for the study.

Exclusion Criteria:

1. Have AJCC Stage IV disease, known distant metastasis, or findings on imaging that are considered to be highly suspicious for distant metastasis.
2. Have injectable tumors impinging upon major airways or blood vessels.
3. Have had prior treatment with recombinant interleukin-12 (IL-12).
4. Have had prior radiation therapy within 28 days for CSCC at the site of injection.
5. Have received live vaccines within 28 days prior to the start of study drug (C1D1).
6. Have any history of transplant-related deoxyribonucleic acid (DNA) viral infections, such as human polyomavirus 1 (BKV), Epstein-Barr virus (EBV), or cytomegalovirus (CMV) within 3 months of C1D1.
7. Have primary or acquired immunodeficient states (e.g., leukemia, lymphoma) requiring active therapy.
8. A WOCBP who has a positive serum pregnancy test prior to C1D1 or female participant who is breastfeeding
9. Have known active uncontrolled hepatitis B, hepatitis C (HCV), or human immunodeficiency virus (HIV) infection.
10. Have active autoimmune disease or medical conditions requiring chronic steroid (i.e., ≥ 20 mg/day prednisone or equivalent) or other immunosuppressive therapy beyond that required for maintenance allograft rejection prevention.
11. Have congestive heart failure, active coronary artery disease, unevaluated new onset angina, unstable angina, or clinically significant cardiac arrhythmias.
12. Have uncontrolled bleeding disorders.
13. Have a history of allergic reactions attributed to compounds of similar biological composition to IL-12, aluminum hydroxide, or drugs formulated with polysorbate-20.
14. Have other systemic conditions or organ abnormalities that may interfere with the conduct the current study.
15. Have any acute or chronic psychiatric problems or substance abuse disorder that make the participant unsuitable for participation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) rate | 3 months
  The percentage of participants who have ≤ 10% viable cancer cells in the surgical pathology sample among all response evaluable participants.

SECONDARY OUTCOMES:
Event Free Survival (EFS) | Up to 3 years
  Time from the first dose of tolododekin alfa to date of event
Relapse Free Survival (RFS) | Up to 3 years
  Time from surgical resection to the earliest date of relapse or death from any cause.
Pathological Complete Response (pCR) | 3 months
  The percentage of participants with complete absence of viable cancer cells in the surgical pathology sample among all response evaluable participants.
Best Overall Response Rate (BORR) | Up to 3 years
  The percentage of participants with a complete response (CR) or partial response (PR) per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 among all response evaluable participants.
Overall Survival (OS) | Up to 3 years
  The time from the administration of tolododekin alfa to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Joe Elassal, MD, MBA, Study Director — Ankyra Therapeutics; Ann Silk, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: No